CLINICAL TRIAL: NCT04833322
Title: Galactose Supplementation for the Treatment of Patients With Mild Malformation of Cortical Development With Oligodendroglial Hyperplasia in Epilepsy (MOGHE): a Pilot Trial
Brief Title: Galactose Supplementation for the Treatment of MOGHE
Acronym: GATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Ruber Internacional (Other)
Responsible Party: Principal Investigator, Angel Aledo-Serrano, Principal Investigator, Hospital Ruber Internacional
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUROLOGIAHRI-01
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Refractory Epilepsy; SLC35A2-CDG - Solute Carrier Family 35 Member A2 Congenital Disorder of Glycosylation
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Galactose

STUDY DESIGN:
Intervention Model Description: Before-and-after pilot clinical trial with a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm group (Experimental): Galactose supplementation
  Interventions: Dietary Supplement: D-Galactose

INTERVENTIONS:
Dietary Supplement: D-Galactose — Galactose supplementation, once per day, up to 1.5g/kg per day

SUMMARY:
Mild malformation of cortical development with oligodendroglial hyperplasia in epilepsy (MOGHE) is a new entity frequently associated with refractory epilepsy and neurodevelopmental disorders. Recently, it has been associated to SLC35A2 (Solute Carrier Family 35 Member A2) brain mosaic pathogenic variants. In addition, patients with germline SLC35A2 pathogenic variants improve with galactose supplementation. Therefore, the investigators aim to elucidate whether d-galactose as an add-on treatment might improve epilepsy and developmental outcomes in patients with MOGHE.

ELIGIBILITY:
Inclusion Criteria:

* MOGHE diagnosis at histopathological examination of the epilepsy surgery tissue.
* Epilepsy refractoriness or ongoing epileptiform activity at EEG.

Exclusion Criteria:

* Allergy to galactose or supplement components.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | 6 months
  Seizure diary
Epileptiform activity at EEG | 6 months
  Epileptiform activity quantification (per epoch)

SECONDARY OUTCOMES:
Behavioral assessment | 6 months
  Teacher and Parent Rating Scale (SNAP-IV) and Conners Continuous Performance Test (CPT-II)
Cognitive assessment | 6 months
  Evaluated with Wechsler Intelligence Scale for Children (WISC-IV) and Behavior Rating Inventory of Executive Function-2 (BRIEF-2)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Aledo-Serrano, MD, PhD, Principal Investigator — Hospital Ruber Internacional
Locations (1):
- Hospital Ruber Internacional, Madrid, Madrid, Comunidad de, Spain

IPD SHARING:
Plan to Share IPD: No